CLINICAL TRIAL: NCT01201265
Title: A Multi Centre, Pilot Phase II Trial Assessing the Efficacy and Safety of Bevacizumab + Gemcitabine + Carboplatin as First Line Treatment for Patients Diagnosed With Triple Negative Metastatic Breast Cancer
Brief Title: A Study of Bevacizumab in Combination With Gemcitabine and Carboplatin in Participants With Triple Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25420
Record Dates: First submitted 2010-09-06; First posted 2010-09-14 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Participants (Experimental): Participants received a combination therapy of bevacizumab with gemcitabine plus carboplatin.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg iv every 3 weeks
  Other Names: Avastin
Drug: Carboplatin — to an AUC = 2, on days 1 and 8 of each 3-week cycle
Drug: Gemcitabine — 1000 mg/m2 iv on days 1 and 8 of each 3-week cycle

SUMMARY:
This multicenter study will assess the efficacy and safety of bevacizumab in combination with gemcitabine and cisplatin as first line treatment in participants with triple negative metastatic breast cancer. Participants will receive bevacizumab at a dose of 15 mg/kg intravenously (iv) every 3 weeks, plus gemcitabine (1000 mg/m2 iv) and carboplatin (iv to an area under curve [AUC]=2) on Days 1 and 8 of each 3-week cycle. Anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, >/= 18 years of age
* Metastatic breast cancer
* Estrogen receptor-, progesterone- and human epidermal growth factor receptor 2 (HER2)-negative disease
* Treatment-naïve for metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematological, renal and liver function
* Patients should have received Anthracyclines and Taxanes in the adjuvant setting
* Women of childbearing potential must agree to use adequate contraception (per institutional standard of care) during treatment and until 6 months after the last administration of investigational products

Exclusion Criteria:

* Prior first line treatment for metastatic breast cancer
* Central nervous system (CNS) metastasis
* Uncontrolled hypertension (> 170/95 mmHg)
* Evidence of bleeding diathesis, coagulopathy or hemorrhage at baseline
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Prior therapy with gemcitabine or carboplatin in the metastatic setting. Participants having received gemcitabine or carboplatin as part of adjuvant therapy are eligible, if recurrence was first documented >6 months after the last exposure to the drug(s)
* Requirement of chronic use of immunosuppressive agents
* HIV, hepatitis B or hepatitis C infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- India (8):
  - Ahmedabad
  - Bangalore
  - Delhi
  - Gandhinagar
  - Mumbai
  - New Delhi
  - Pune
  - Vellore

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants received a combination therapy of bevacizumab 15 milligram per kilogram (mg/kg) intravenous every 3 weeks with carboplatin recommended dose (area under curve [AUC]= 2) along with gemcitabine 1000 mg/ metre square (m^2) on days 1 and 8 of each 3 week cycle.
Period: Overall Study
Arm/Group | All Participants
Started | 40
Completed | 2
Not Completed | 38
Not completed — Death | 14
Not completed — Insufficient Therapeutic Response | 3
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 7
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) was calculated in days from the date of registration until the earliest date of documented disease progression or death. The median PFS time with 95% confidence interval (CI) was estimated using Kaplan Meier method. The progression-free survival was assessed utilizing computer tomography (CT)/ magnetic resonance imaging (MRI)/bone scans and X-ray and Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1. Progression of disease is defined as at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: From the date of registration until the disease progression or death (up to 1541 days).
Population: Efficacy analysis population included all participants who received at least one dose of study treatment and with at least one efficacy assessment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 40
days | 255 [157 to 465]

2. Secondary Outcome: Percentage of Participants Achieving an Overall Response
Description: The overall response rate (ORR) was defined as complete response (CR) + partial response (PR). ORR was summarized using number and percentage along with two-sided 95% Pearson-Clopper CI. The overall response rate was assessed utilizing the RECIST v. 1.1. CR: disappearance of all target and non-target lesions (TLs) and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 millimeter (mm). PR: at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of diameters.
Time Frame: From the date of registration until the disease progression or death (up to 1541 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
percentage of participants | 50.0 [33.8 to 66.2]

3. Secondary Outcome: Percentage of Participants Achieving a Clinical Benefit Response (CBR)
Description: Clinical benefit response was defined as a complete response (CR), partial response (PR) or stable disease (SD). CBR was assessed using Recist v.1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of registration until the disease progression or death (up to 1541 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
percentage of participants | 92.5 [79.6 to 98.4]

4. Secondary Outcome: Time to Progression (TTP)
Description: Duration of time to progression (TTP) was estimated using the Kaplan-Meier method. The time to progression was calculated in days from the date of registration until the earliest date of documented disease progression.
Time Frame: From the date of registration until the disease progression (up to 1541 days).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 40
days | 269.0 [182.0 to 551.0]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the date of the first study drug dose to the date of death from any cause. The median overall survival time with 95%CI was estimated using Kaplan-Meier method.
Time Frame: From the date of registration until the disease progression or death (up to 1541 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 40
days | 475.0 [358.0 to 759.0]

6. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 28 days after termination of study treatment (approximately 1569 days)
Population: Safety population included all participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
participants | 24

7. Secondary Outcome: Change From Baseline to Cycle 6 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30)
Description: The EORTC QLQ-C30 (version 3.0) questionnaire incorporates 9 multi scale items: 5 functional scales (physical, role, cognitive, emotional and social); 3 symptom scales (fatigue, pain and nausea & vomiting); and a global health and quality-of-life scale. It contains 30 questions. The score for each item and the overall score ranges from 0 to 100. A high overall scale and subscale scores represent improved health status. However, in case of symptoms, higher scores suggest increased perception of these symptoms.
Time Frame: Baseline, cycle 6
Population: Efficacy analysis population included all participants who received at least one dose of study treatment and with at least one efficacy assessment. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 40
units on a scale
  Baseline; physical (n=40) | 69.33 (20.963)
  Change at Cycle 6; physical (n=28) | -8.82 (24.154)
  Baseline; role (n=40) | 71.26 (25.311)
  Change at Cycle 6; role (n=28) | -5.36 (22.705)
  Baseline; cognitive (n=40) | 74.58 (24.745)
  Change at Cycle 6; cognitive (n=28) | -4.17 (27.444)
  Baseline; emotional (n=40) | 61.87 (22.396)
  Change at Cycle 6; emotional (n=28) | -15.78 (23.929)
  Baseline; social (n=40) | 65.42 (29.330)
  Change at Cycle 6; social (n=28) | -8.33 (27.026)
  Baseline; fatigue (n=40) | 42.21 (20.026)
  Change at Cycle 6; fatigue (n=28) | 8.35 (25.785)
  Baseline; pain (n=40) | 34.58 (25.428)
  Change at Cycle 6; pain (n=28) | 13.09 (33.744)
  Baseline; nausea and vomiting (n=40) | 16.67 (20.326)
  Change at Cycle 6; nausea and vomiting (n=28) | 2.38 (19.082)
  Baseline; global health & QOL (n=40) | 58.55 (17.750)
  Change at Cycle 6; global health & QOL (n=28) | -3.86 (17.191)

8. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Change from baseline in SBP was analyzed by overall response (CR+PR, SD+PD).
Time Frame: Baseline, Cycle 6, 12 of treatment
Population: Safety population included all participants who received at least one dose of study treatment. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | All Participants
Number analyzed (Participants) | 40
millimetre of mercury (mmHg)
  Baseline; CR+PR (n= 19) | 124.8 (12.86)
  Change at cycle 6; CR+PR (n=14) | -4.6 (12.16)
  Change at cycle 12; CR+PR at cycle 12 (n=5) | -4.0 (18.17)
  Baseline; SD+PD (n= 18) | 123.6 (6.82)
  Change at cycle 6; SD+PD at cycle 6 (n=13) | 0.2 (12.68)
  Change at cycle 12; SD+PD at cycle 12 (n=4) | -6.3 (17.97)

9. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: Change from baseline in DBP was analyzed by overall response (CR+PR, SD+PD).
Time Frame: Baseline, Cycle 6, 12 of treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 40
mmHg
  Baseline; CR+PR (n= 19) | 80.4 (9.65)
  Change at cycle 6; CR+PR (n=14) | -4.1 (10.83)
  Change at cycle 12; CR+PR (n=5) | -2.0 (14.83)
  Baseline; SD+PD (n= 18) | 78.9 (7.58)
  Change at cycle 6; SD+PD (n=13) | 2.3 (10.92)
  Change at cycle 12; SD+PD (n=4) | 7.5 (12.58)

ADVERSE EVENTS:
Time Frame: Up to 28 days after termination of study treatment (approximately 1569 days)
Groups:
- All Particiapants: Participants received a combination therapy of bevacizumab 15 milligram per kilogram (mg/kg) intravenous every 3 weeks with carboplatin recommended dose (area under curve [AUC]= 2) along with gemcitabine 1000 mg/ metre square (m^2) on days 1 and 8 of each 3 week cycle.
Arm/Group | All Particiapants
Serious Adverse Events (participants affected / at risk) | 17/40
Other Adverse Events (participants affected / at risk) | 18/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Particiapants (N=40)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Pericardial Effusion (Cardiac disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Disease Progression (General disorders) | 6
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 3
Septic Shock (Infections and infestations) | 1
Streptococcal Infection (Infections and infestations) | 1
Viral Respiratory Tract Infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Oxygen Saturation Decreased (Investigations) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Particiapants (N=40)
Anaemia (Blood and lymphatic system disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Stomatitis (Gastrointestinal disorders) | 2
Disease Progression (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.